CLINICAL TRIAL: NCT07024810
Title: Effect of Nurse-assessed Remote Ischemic Preconditioning on Improving Exercise Capacity, Endothelial Function, and Arterial Stiffness in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: PIRIC-FEp Stud
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG: 2025/PI0625
Record Dates: First submitted 2025-05-30; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: HF - Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic preconditioning (Experimental): Participants randomized to the PIR intervention group will receive a hand-held blood pressure device (Welch Allyn DuraShock™ DS45, NY, USA) to self-administer PIR. The cuff will be placed around the upper arm and inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, and this cycle will be repeated another three times. This process will be performed 5 days a week for 3 months.
  Interventions: Other: remote ischemic preconditioning
- normal routine and to refrain from any new physical activity or change in eating habits. (No Intervention)

INTERVENTIONS:
Other: remote ischemic preconditioning — Participants randomized to the PIR intervention group will receive a hand-held blood pressure device (Welch Allyn DuraShock™ DS45, NY, USA) to self-administer PIR. The cuff will be placed around the upper arm and inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, and this cycle will be repeated another three times. This process will be performed 5 days a week for 3 months. The arm on which participants will apply the PIR is the left arm. Participants will be supervised during their first PIR session and every 15 days to ensure that it is performed correctly and, they will be free to perform the PIR at any time during the day and will record it in a diary to monitor compliance. Participants will be instructed to follow their normal routine and refrain from engaging in any new physical activity or changing their eating habits.
  Arms: remote ischemic preconditioning

SUMMARY:
The PIRIC-FEp study will be a randomized clinical trial in sedentary patients with heart failure and stable preserved ejection fraction.

Objectives: 1) To evaluate the efficacy of remote ischemic preconditioning performed by nurses, a noninvasive cardioprotective intervention that uses cycles of ischemia and reperfusion in the extremities, in improving exercise capacity, cardiac function, endothelial function and arterial stiffness, and 2) To analyze its impact on quality of life and its cost-effectiveness compared to conventional treatment.

Methodology: Patients will be recruited in Health Centers in the city. Those assigned to the intervention group will wear a self-administered blood pressure cuff, inflated to 220 mmHg for 5 minutes, followed by 5 minutes of deflation, in repeated cycles four times, five days a week for three months. The control group will receive standard counseling. All participants will be examined, at baseline and at three months. Adherence will be defined as completing at least 70% of the sessions. Different parameters will be evaluated, including sociodemographic variables, patient's medical history, echocardiography, cardiopulmonary exercise test, endothelial function, arterial stiffness, quality of life, spirometry, blood tests, among others. The study will be approved by an Ethics Committee, participants will be informed and will have to sign a written consent. The statistical analysis will include three phases: verification of randomization, use of covariance models for dependent variables, and sensitivity analysis with propensity score matching. All analyses will be performed on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

1. HF-PEF (diagnosis according to the ESC 2021 criteria)

   1. Signs and symptoms of HF
   2. A left ventricular ejection fraction ≥50%.
   3. Objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of left ventricular diastolic dysfunction/elevated left ventricular filling pressures, including elevated natriuretic peptides
2. Sedentary men and women (structured exercise <2 x 30 min/week).
3. Age ≥40 years
4. Written informed consent
5. Clinically stable for 6 weeks
6. Optimal medical treatment for ≥6 weeks.

Exclusion Criteria:

1. Non-cardiac causes of HF symptoms:

   * Significant valvular or coronary artery disease
   * Uncontrolled hypertension or arrhythmias
   * Primary cardiomyopathies
2. Significant pulmonary disease (FEV1<50% predicted, GOLD III-IV)
3. Inability to exercise or conditions that may interfere with exercise intervention.
4. Myocardial infarction within the last 3 months.
5. Patients with diabetes and/or peripheral vascular disease.
6. Signs of ischemia during maximal cardiopulmonary stress test.
7. Comorbidity that may influence prognosis at one year.
8. Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | From enrollment to the end of treatment at 12 weeks
  The 6-minute walking test will be performed in a 30-meter corridor, which will be carried out by walking back and forth along this section, which will be delimited by cone-type indicators. These signs shall be placed at a distance of 29 meters from each other, leaving 0.5 meters at each end for the subject to turn. The test shall be performed accompanied by the examiner.
  Unit of measure: Meters. Interpretation: Higher values indicate better exercise capacity.
Endothelial function | From enrollment to the end of treatment at 12 weeks
  Carotid intima-media layer thickness: by ultrasound with the Sonosite SII device (Sonosite Inc., Bothell, Washington, USA).
  Unit of Measure: Millimeters (mm) Interpretation: Lower values indicate better endothelial function.
Pulse wave velocity (PWV) | From enrollment to the end of treatment at 12 weeks
  Arterial stiffness will be assessed using the SphygmoCor System to calculate carotid-femoral pulse wave velocity.
  Unit of Measure: Meters per second (m/s) Interpretation: Lower values indicate better arterial elasticity.
Radial augmentation index (rAIx) | From enrollment to the end of treatment at 12 weeks
  The radial augmentation index will be calculated using the SphygmoCor System. Formula: (SBP2 - DBP)/(SBP - DBP) x 100 (%).
  Unit of Measure: Percentage (%) Interpretation: Lower values indicate better vascular function.
Central augmentation index (cAIx) | From enrollment to the end of treatment at 12 weeks
  The central augmentation index will be calculated using the SphygmoCor System. Formula: Central pulse pressure increase x 100 / Pulse pressure.
  Unit of Measure: Percentage (%) Interpretation: Lower values indicate better vascular function.

SECONDARY OUTCOMES:
Body weight | From enrollment to the end of treatment at 12 weeks
  Weight will be assessed using a Seca® 861 digital scale. The mean of two measurements will be recorded, with participants barefoot and wearing light clothing.
  Unit of Measure: Kilograms (kg) Interpretation: Lower weight may indicate a reduction in overall adiposity depending on context.
Height | From enrollment to the end of treatment at 12 weeks
  Height will be measured using a wall-mounted stadiometer (Seca® 222). The mean of two measurements will be recorded with participants barefoot, in upright position.
  Unit of Measure: Meters (m) Interpretation: Stable in adults; used to calculate BMI.
Body mass index (BMI) | From enrollment to the end of treatment at 12 weeks
  BMI will be calculated as weight in kilograms divided by the square of height in meters (kg/m²).
  Unit of Measure: kg/m² Interpretation: Lower values generally indicate lower body fat in the absence of muscle mass loss.
Waist circumference | From enrollment to the end of treatment at 12 weeks
  Waist circumference will be measured with a flexible tape at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, at the end of a normal exhalation. The average of three measurements will be used.
  Unit of Measure: Centimeters (cm) Interpretation: Lower values suggest reduced central adiposity.
Body fat percentage | From enrollment to the end of treatment at 12 weeks
  Body fat percentage will be assessed using an 8-electrode bioelectrical impedance analyzer (Tanita® BC-418 MA). The mean of two measurements will be recorded.
  Unit of Measure: Percentage (%) Interpretation: Lower values may indicate improved body composition.
Systolic blood pressure (SBP) | From enrollment to the end of treatment at 12 week
  Systolic blood pressure will be measured as the mean of two readings separated by 5 minutes. Measurements will be taken in a seated position using the Omron® H907 monitor.
  Unit of Measure: Millimeters of mercury (mmHg) Interpretation: Lower SBP indicates improved cardiovascular function.
Diastolic blood pressure (DBP) | From enrollment to the end of treatment at 12 weeks
  Diastolic blood pressure will be measured as the mean of two readings separated by 5 minutes, using the same protocol and device as for SBP.
  Unit of Measure: Millimeters of mercury (mmHg) Interpretation: Lower DBP indicates improved cardiovascular function.
Grip strength | From enrollment to the end of treatment at 12 weeks
  Muscular strength will be assessed using the TKK 5401 Grip-D dynamometer (Takey®, Tokyo, Japan). Manual grip force will be recorded in kilograms.
  Unit of Measure: Kilograms (kg) Interpretation: Higher grip strength reflects better muscular function.
Step rate (cadence) | From enrollment to the end of treatment at 12 weeks
  The average number of steps per minute will be monitored using the Fitbit Inspire 3 over a continuous 9-day period.
  Unit of Measure: Steps per minute Interpretation: Higher cadence indicates greater physical activity.
Heart rate | From enrollment to the end of treatment at 12 weeks
  Mean heart rate will be continuously recorded in 1-minute intervals using the Fitbit Inspire 3 for 9 consecutive days.
  Unit of Measure: Beats per minute (bpm) Interpretation: Lower resting heart rate may indicate improved cardiovascular fitness.
Sleep duration | From enrollment to the end of treatment at 12 weeks
  Daily sleep duration (in hours) will be recorded using the Fitbit Inspire 3 over a 9-day period.
  Unit of Measure: Hours per night Interpretation: Longer sleep duration (within healthy ranges) is generally favorable.
Sleep quality score | From enrollment to the end of treatment at 12 weeks
  Sleep quality will be estimated using proprietary algorithms from the Fitbit Inspire 3, generating a composite sleep score based on movement, interruptions, and time spent in sleep stages.
  Unit of Measure: Units on a 0-100 scale Interpretation: Higher scores represent better sleep quality.
Metabolic equivalents (METs) | From enrollment to the end of treatment at 12 weeks
  METs will be estimated based on movement and heart rate using the Fitbit Inspire 3, representing energy expenditure relative to rest.
  Unit of Measure: METs Interpretation: Higher METs indicate more intense or sustained physical activity.
DNA sample collection for genotyping | Baseline mesaurements
  Saliva samples (1-3 mL) will be collected in sterile tubes with a preservation reagent to maintain DNA integrity. Samples will be used for genotyping analysis.
  Unit of Measure: Presence or absence of adequate sample for genotyping (Yes/No) Interpretation: Successful collection enables subsequent genetic analysis; no scoring or numerical outcome applies.
Physical activity level (IPAQ total MET-min/week) | From enrollment to the end of treatment at 12 weeks
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). It categorizes activity levels as low, moderate, or high, and estimates total weekly energy expenditure in MET-minutes.
  Unit of Measure: MET-minutes per week Interpretation: Higher values indicate greater total physical activity.
Physical fitness self-perception (IFIS total score) | From enrollment to the end of treatment at 12 weeks
  Physical fitness will be assessed using the International Fitness Scale (IFIS), a validated self-report questionnaire evaluating five components: general fitness, cardiorespiratory fitness, muscular strength, speed-agility, and flexibility. Each item is scored on a 5-point Likert scale (1 = very poor, 5 = very good).
  Unit of Measure: Score (1-5 for each item, or total score range: 5-25) Interpretation: Higher scores indicate better perceived physical fitness.
Adherence to the Mediterranean diet (MEDAS-14 total score) | From enrollment to the end of treatment at 12 weeks
  Adherence to the Mediterranean diet will be assessed using the 14-item Mediterranean Diet Adherence Screener (MEDAS-14). Each item is scored as 0 or 1, resulting in a total score ranging from 0 to 14.
  Unit of Measure: Score (0-14) Interpretation: Higher scores indicate greater adherence to the Mediterranean dietary pattern.
Health-related quality of life (SF-12 total score) | From enrollment to the end of treatment at 12 weeks
  The 12-item Short Form Health Survey (SF-12) will be used to assess general quality of life. It includes two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each score ranges from 0 to 100, with higher scores indicating better health status.
  Unit of Measure: Score (0-100 for each component) Interpretation: Higher scores represent better perceived physical and mental health.
Heart failure-related quality of life (MLWHFQ total score) | From enrollment to the end of treatment at 12 weeks
  The Minnesota Living With Heart Failure Questionnaire (MLWHFQ) evaluates the impact of heart failure on patients' quality of life. It contains 21 items rated from 0 (no impact) to 5 (very much), resulting in a total score ranging from 0 to 105.
  Unit of Measure: Score (0-105) Interpretation: Lower scores indicate better quality of life and fewer symptoms related to heart failure.
Consumption of highly processed foods (SQ-HPF total score) | From enrollment to the end of treatment at 12 weeks
  The frequency and quantity of consumption of highly processed foods will be assessed using the Short Questionnaire for the Assessment of Highly Processed Food Consumption (SQ-HPF). The questionnaire includes 14 food categories, each scored based on consumption frequency. The total score ranges from 0 to 28.
  Unit of Measure: Score (0-28) Interpretation: Higher scores indicate more frequent consumption of highly processed foods.
Fasting glucose | From enrollment to the end of treatment at 12 weeks
  Fasting plasma glucose will be measured using the Roche Diagnostics® Cobas 8000 system.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Lower levels indicate better glycemic control.
Total cholesterol | From enrollment to the end of treatment at 12 weeks
  Serum total cholesterol will be analyzed on the Roche Diagnostics® Cobas 8000 platform.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Lower levels generally reflect better lipid profile.
Triglycerides | From enrollment to the end of treatment at 12 weeks
  Serum triglycerides will be measured using the Roche Diagnostics® Cobas 8000 system.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Lower values are associated with improved metabolic health.
HDL cholesterol | From enrollment to the end of treatment at 12 weeks
  High-density lipoprotein cholesterol will be assessed via the Cobas 8000 system.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Higher values are considered cardioprotective.
LDL cholesterol | From enrollment to the end of treatment at 12 weeks
  Low-density lipoprotein cholesterol will be measured using the Roche Cobas 8000 analyzer.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Lower values reduce cardiovascular risk.
Apolipoprotein A1 | From enrollment to the end of treatment at 12 weeks
  Apolipoprotein A1 will be determined with the Roche Diagnostics® Cobas 8000 system.
  Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Higher levels are associated with better HDL function.
Apolipoprotein B | From enrollment to the end of treatment at 12 weeks
  Apolipoprotein B levels will be measured using the Cobas 8000 platform. Unit of Measure: Milligrams per deciliter (mg/dL) Interpretation: Lower values are associated with reduced atherogenic risk.
Fasting insulin | From enrollment to the end of treatment at 12 weeks
  Insulin concentration will be measured using the Abbott® Architect platform. Unit of Measure: Micro-international units per milliliter (µIU/mL) Interpretation: Lower fasting insulin suggests better insulin sensitivity.
High-sensitivity C-reactive protein (hs-CRP) | From enrollment to the end of treatment at 12 weeks
  Serum hs-CRP will be assessed using the Roche Cobas 8000 system. Unit of Measure: Milligrams per liter (mg/L) Interpretation: Lower levels reflect lower systemic inflammation.
Glycated hemoglobin (HbA1c) | From enrollment to the end of treatment at 12 weeks
  HbA1c will be determined using high-performance liquid chromatography (HPLC) on the ADAMS A1c HA-8180V analyzer (A. Menarini Diagnostics®), NGSP-certified method.
  Unit of Measure: Percentage (%) Interpretation: Lower values indicate improved long-term glycemic control.

IPD SHARING:
Plan to Share IPD: Yes